CLINICAL TRIAL: NCT06547229
Title: Clinicopathological Features and Genetic Susceptibility Screening of Recurrent Drug-induced Liver Injury
Acronym: RDILI-GS
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Xinyan, Professor, Beijing Friendship Hospital
Other Study IDs: 2024-P2-238
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Drug-induced Liver Injury
Keywords: Genetic Susceptibility; HLA; Endpoint Event(s); Drug-induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Retrospective and Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to screening for clinical, pathological and HLA features in patients with recurrent drug-induced liver injury. The main question it aims to answer is: Which patients with drug-induced liver injury need to be more cautious when re-dosing?

DETAILED DESCRIPTION:
Research Objectives:

1. To summarise the clinicopathological characteristics of patients with recurrent drug-induced liver injury (DILI) in the Liver Disease Centre of Beijing Friendship Hospital in the past 10 years.
2. Compare the differences in clinicopathological characteristics between patients with only one episode of different drug use and those with recurrent DILI, and predict the risk/protective factors in patients with recurrent DILI.
3. Explore the susceptibility genes in patients with recurrent DILI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for recurrent drug induced liver injury:

  1. Liver enzymes returns to normal or has a tendency to remission after the first drug liver injury;
  2. Signs and symptoms of liver injury after the patient takes the different drugs for liver injury again, and the liver enzymes returns to normal through follow-up.

Inclusion criteria for drug induced liver injury:

1. RUCAM ≥6 and met one of the following biochemical conditions: (1)ALT≥5 ULN, (2) or ALP ≥2 ULN, (3) or ALT≥3 ULN and TBil≥2 ULN.
2. RUCAM between 3-5, five experienced hepatologists in leading site evaluate and vote the diagnosis of DILI, the case would be enrolled if only ≥4 out of 5 hepatologists agree with the diagnosis.
3. Onset to enrollment ≤3 months.

Exclusion Criteria:

* 1. Hepatotropic viral infection: hepatitis A, B, C, D and E. 2. Non-hepatotropic viral infection: cytomegalovirus (CMV) and Epstein-Barr virus (EBV), etc.

  3. Hypoxic ischemic hepatitis and congestive liver disease. 4. Alcohol consumption: male >40g/d, female >20g/d, and ≥5 years.5. Biliary obstruction, primary biliary cholangitis; primary sclerosing cholangitis.

  6. Autoimmune hepatitis: International Autoimmune Hepatitis Group (IAHG)simplified score ≥6 or complicated score ≥10, or differentiation from autoimmune hepatitis is impossible during enrollment.

  7. Parasitic infection. 8. Sepsis. 9. Previous liver transplantation or bone marrow transplantation. 10. Pregnancy or lactation. 11. Genetic and metabolic liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with recurrent drug-induced liver injury
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Death/Liver transplantation | 1 year
  DILI has a primary, contributory role for the death (liver-related mortality) or no role for the death (all-cause mortality) .
  DILI is the primary indication for liver transplantation.
Acute Liver Failure | 1 year
  Acute liver failure is defined as elevated bilirubin and prolonged international normalized ratio (INR) ≥1.5 accompaniedby mental disturbance within 26 weeks after DILI onset without underlying chronic liver diseases.
Recovery | 1 year
  Recovery status is defined as clinical and biochemical resolution within 1 year after DILI onset, with alanineaminotransferase (ALT) or aspartate aminotransferase (AST) ≤40 U/L, alkaline phosphatase (ALP) ≤150 U/L, and totalbilirubin (TB) ≤1.5 upper limits of normal (ULN) (25.65 μmol/L).

SECONDARY OUTCOMES:
chronic DILI | 2 years
  Chronicity is defined as the presence of any one of the following: (i) persistently elevated liver biochemistry indexes; (ii)radiological or histological evidence of persistent liver injury at one year after DILI onset.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan Zhao, Study Chair — Beijing Friendship Hospital
Locations (1):
- Liver Research Center, Beijing Friendship Hospital, Key Laboratory on Translational Medicine on Cirrhosis, National Clinical Research Center for Digestive Disease, Capital Medical University, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No